CLINICAL TRIAL: NCT03006822
Title: Time Effect of the Pressure Release Technique Application in the Latent Myofascial Trigger Points of the Levator Scapulae
Brief Title: Time Effect of the Pressure Release Technique Application in the Latent Myofascial Trigger Points
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Prof. Dr. Daniel Pecos Martín, Dr. Pecos-Martin, Daniel (Principal Investigator), University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Universidad de Alcalá
Record Dates: First submitted 2016-10-27; First posted 2016-12-30 (Estimated); Last update posted 2017-10-04 (Actual); Status verified 2017-10

CONDITIONS: Myofascial Pain Syndrome
Keywords: Myofascial Trigger Points; Liberation for Pression; Therapy Soft Tissue
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Application 90 minutes pressure release (Experimental): Subjects will receive a pressure release technique for 90 seconds in the levator scapula muscle
  Interventions: Other: Pressure release 90
- Application 60 minutes pressure release (Experimental): Subjects will receive a pressure release technique for 60 seconds in the levator scapula muscle
  Interventions: Other: Pressure release 60
- Application 30 minutes pressure release (Experimental): Subjects will receive a pressure release technique for 30 seconds in the levator scapula muscle
  Interventions: Other: Pressure release 30

INTERVENTIONS:
Other: Pressure release 90 — This is a massage technique that aims is eliminate myofascial trigger points for to treat muscle pain.
  Other Names: soft tissue massage; Compression ischemic massage technique
  Arms: Application 90 minutes pressure release
Other: Pressure release 60 — This is a massage technique that aims is eliminate myofascial trigger points for to treat muscle pain.
  Other Names: Compression ischemic massage technique; soft tissue massage
  Arms: Application 60 minutes pressure release
Other: Pressure release 30 — This is a massage technique that aims is eliminate myofascial trigger points for to treat muscle pain.
  Other Names: Compression ischemic massage technique; soft tissue massage
  Arms: Application 30 minutes pressure release

SUMMARY:
Background: Latent myofascial trigger points (MTrPs) of the levator scapulae are high prevalent and may influence the neck and shoulder conditions. The pressure release is one of the most recommended manual therapy techniques.

Objective: To determine the time effect of the pressure release technique application in the latent MTrPs of the levator scapulae muscle.

Design: A three-arm (1:1:1 ratio), double-blinded, parallel, randomized clinical trial.

The manual technique than us apply, be sustained digital pressure with thumbs or with the 2nd-3rd fingers on the PGM below the pain threshold and gradually increases up to a ceiling of tissue resistance (barrier), as decreases, adds more pressure. different times of sustained pressure and the number of repetitions depending on time 30 (group 1, acts as a control), 60 (group 2) and 90 seconds (group 3) shall apply.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with aged between 18 and 60 years.
* Subjects with presence of latent PGM levator scapulae muscle.

Exclusion Criteria:

* Pregnant.
* Subjects with spontaneous pain.
* Subjects with neck or shoulder pain.
* Subjects with musculoskeletal injuries.
* Subjects with neurological problems.
* Fibromyalgia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2017-03-20 (Actual); Study Completion 2017-07-10 (Actual)

PRIMARY OUTCOMES:
Pain pressure threshold (PPT) | Change from Baseline PPT at one week
  PPT is defined as the minimal amount of pressure that produce pain. The investigators will measure the muscle levator scapular tenderness.

SECONDARY OUTCOMES:
Strength muscle | Change from Baseline strength muscle at one week
  The investigators will measure strength muscle with a handheld dynamometer. the subject will have to perform a movement of cervical extension resistance against.

OTHER OUTCOMES:
Range of cervical mobility | Change from Baseline range of cervical mobility at one week
  The range of cervical mobility will has measure with cervical goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Pecos-Martin, Doctor, Study Director — Alcalá University (Physical Therapy and pain group)
Locations (1):
- Grupo Fisioterapia y Dolor, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pecos-Martin D, Ponce-Castro MJ, Jimenez-Rejano JJ, Nunez-Nagy S, Calvo-Lobo C, Gallego-Izquierdo T. Immediate effects of variable durations of pressure release technique on latent myofascial trigger points of the levator scapulae: a double-blinded randomised clinical trial. Acupunct Med. 2019 Jun;37(3):141-150. doi: 10.1136/acupmed-2018-011738. Epub 2019 May 7. PMID 31060367